CLINICAL TRIAL: NCT01126359
Title: Lidocaine Analgesia For Removal Of Wound Vacuum Assisted Closure Dressings: A Randomized Double Blinded Controlled Trial
Brief Title: Lidocaine Analgesia For Removal Of Wound Vac Dressings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Eric Kubiak, M.D., University of Utah
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 29398
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Results first posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Pain
Keywords: Wound Vacuum Assisted Dressings; Lidocaine; Dressing change; Pain management; palliative care
MeSH Terms: conditions — Pain; Agnosia | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine then Placebo-Saline (Placebo Comparator)
  Interventions: Drug: Lidocaine; Drug: Placebo-Saline
- Placebo-Saline then Lidocaine (Active Comparator)
  Interventions: Drug: Lidocaine; Drug: Placebo-Saline

INTERVENTIONS:
Drug: Lidocaine — Interventional dressing change: iv or po pain medication with injection of 1% lidocaine retrograde up the suction tube into the sponge.
  Other Names: xylocaine
Drug: Placebo-Saline — Control dressing change: iv or po pain medication and injection of 0.9% normal saline retrograde up the suction tube.
  Other Names: 0.9% normal saline

SUMMARY:
The purpose of this prospective study is to compare pain levels and pain medication dose requirements in patients with topical negative pressure (TNP) dressings removed in a standard manner (i.v. or p.o. pain meds) compared to dressings removed with lidocaine analgesia, via injection retrograde up the suction tube into the foam prior to removal. Our null hypothesis is that there will be no difference in overall pain scores or medication requirements when patients receive a saline, control injection and pain medications, compared to when their dressings are changed with a lidocaine injection into the sponge, with pain medications. Our objective is to disprove this null hypothesis with statistical significance.

ELIGIBILITY:
Inclusion Criteria:

1. wounds to which a split-thickness autologous skin graft applied;
2. infected wounds after debridement;
3. open fracture wounds;
4. acute soft-tissue wounds (with exposed tendon, bone, hardware, and/or joint);
5. fasciotomy wounds after compartment syndrome;
6. chronic non-healing wounds;
7. surgical wounds that are difficult to close due to tension; or
8. wounds with external fixation pins or tubes with irritation or drainage.

Exclusion Criteria:

1. allergy to lidocaine;
2. allergy to the polyurethane foam or impermeable seal;
3. malignancy associated with the wound;
4. extremity insensate to pain due to any cause (including diabetic neuropathy, or any neurologic disorder therein);
5. pregnancy as diagnosed by urine pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik N Kubiak, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Webb LX. New techniques in wound management: vacuum-assisted wound closure. J Am Acad Orthop Surg. 2002 Sep-Oct;10(5):303-11. doi: 10.5435/00124635-200209000-00002. PMID 12374481
- [Background] Garner GB, Ware DN, Cocanour CS, Duke JH, McKinley BA, Kozar RA, Moore FA. Vacuum-assisted wound closure provides early fascial reapproximation in trauma patients with open abdomens. Am J Surg. 2001 Dec;182(6):630-8. doi: 10.1016/s0002-9610(01)00786-3. PMID 11839329
- [Background] Choe JH, Kwak KW, Hong JH, Lee HM. Efficacy of lidocaine spray as topical anesthesia for outpatient rigid cystoscopy in women: a prospective, randomized, double-blind trial. Urology. 2008 Apr;71(4):561-6. doi: 10.1016/j.urology.2007.11.057. Epub 2008 Feb 15. PMID 18279921
- [Result] Christensen TJ, Thorum T, Kubiak EN. Lidocaine analgesia for removal of wound vacuum-assisted closure dressings: a randomized double-blinded placebo-controlled trial. J Orthop Trauma. 2013 Feb;27(2):107-12. doi: 10.1097/BOT.0b013e318251219c. PMID 23343829

RESULTS

PARTICIPANT FLOW:
Groups:
- Lidocaine Then Placebo-Saline: Interventional dressing change: iv or po pain medication with injection of 1% lidocaine retrograde up the suction tube into the sponge. Then, control dressing change: iv or po pain medication and injection of 1% saline retrograde up the suction tube.
- Placebo-Saline Then Lidocaine: Control dressing change: iv or po pain medication and injection of 1% saline retrograde up the suction tube. Then, interventional dressing change: iv or po pain medication with injection of 1% lidocaine retrograde up the suction tube into the sponge.
Period: First Intervention (20-minutes)
Arm/Group | Lidocaine Then Placebo-Saline | Placebo-Saline Then Lidocaine
Started | 5 | 6
Completed | 5 | 5
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Dressing Replacement/Healing (48-hours)
Arm/Group | Lidocaine Then Placebo-Saline | Placebo-Saline Then Lidocaine
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention (20-minutes)
Arm/Group | Lidocaine Then Placebo-Saline | Placebo-Saline Then Lidocaine
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes participants randomized to receive Lidocaine first, then Placebo-Saline; and vice versa.
Arm/Group | All Study Participants
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale Pain Score
Description: Visial Analog Pain Scores (VAS) range from 0 (no pain) - 10 (worst pain ever). Visial Analog Pain Scores are determined at each pain measurement time point (during/after VAC dressing removal).
Time Frame: 20 minutes
Measure: Mean (95% Confidence Interval); unit: Visial Analog Pain Score (VAS)
Groups:
- Lidocaine: All patients who received lidocaine prior to VAC dressing change.
- Placebo-Saline: All patients who received placebo-saline prior to VAC dressing change.
- Lidocaine Minus Placebo-Saline Difference: Includes participants randomized to receive Lidocaine first, then Placebo-Saline; and vice versa. Visial Analog Pain Scores are determined at each pain measurement time point (during/after VAC dressing removal) as the Lidocaine minus Placebo-Saline VAS difference for each participant. A negative VAS difference indicates a reduction in the level of pain with Lidocaine compared to Placebo-Saline utilizing crossover intervention.
Arm/Group | Lidocaine | Placebo-Saline | Lidocaine Minus Placebo-Saline Difference
Number analyzed (Participants) | 10 | 11 | 11
Visial Analog Pain Score (VAS)
  During VAC change | 6.5 [5.5 to 7.4] | 8.9 [8.0 to 9.7] | -2.4 [-3.0 to -1.7]
  5 min post-VAC change | 4.4 [3.2 to 5.7] | 6.4 [5.3 to 7.5] | -2.0 [-3.3 to -0.8]
  10 min post VAC change | 3.2 [2.0 to 4.5] | 4.7 [3.6 to 5.8] | -1.5 [-2.8 to -0.1]
  20 min post VAC change | 2.4 [1.3 to 3.5] | 4.2 [3.2 to 5.1] | -1.8 [-3.0 to -0.6]

2. Secondary Outcome: Break-through Narcotic Requirement
Description: Patient break-through narcotic requirements in morphine equivalents are 0.2 mg of dilaudid = 1 mg of morphine, iv., used during and after VAC dressing change.
Time Frame: 20 minutes
Measure: Mean (95% Confidence Interval); unit: Narcotic Requirements (mg)
Groups:
- Lidocaine Minus Placebo-Saline Difference: Includes participants randomized to receive Lidocaine first, then Placebo-Saline; and vice versa. Each patient narcotic requirements are determined at each measured time point (during/after VAC dressing removal) as the Lidocaine minus Placebo-Saline difference (mg). A negative narcotic requirement difference indicates a reduction in medication dosed (mg) used during and after VAC dressing change in a crossover intervention technique.
Arm/Group | Lidocaine | Placebo-Saline | Lidocaine Minus Placebo-Saline Difference
Number analyzed (Participants) | 10 | 11 | 11
Narcotic Requirements (mg)
  During VAC change | 1.3 [0.2 to 2.3] | 3.0 [2.0 to 3.9] | -1.7 [-2.3 to -1.1]
  5 min post-VAC change | 0.8 [0.0 to 1.6] | 1.1 [0.4 to 1.9] | -0.4 [-1.0 to -0.2]
  10 min post VAC change | 0.2 [-0.3 to 0.6] | 0.4 [0.0 to 0.8] | -0.2 [-0.8 to 0.4]
  20 min post VAC change | 0.0 [-0.4 to 0.3] | 0.3 [0.0 to 0.6] | -0.3 [-0.7 to 0.1]

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | First Intervention (Lidocaine) | First Intervention (Placebo) | Second Intervention (Placebo) | Second Intervention (Lidocaine)
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Overall subjectivity of pain and dosing of narcotic medications, all male cohort, timing of wound VAC changes, did not define the ideal lidocaine dosing for VAC changes or dosing method.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes